CLINICAL TRIAL: NCT05331911
Title: Impact of Propofol-Based Total Intravenous Anesthesia Versus Anesthesia With Sevoflurane
Brief Title: Impact of Propofol-Based Total Intravenous Anesthesia Versus Anesthesia With Sevoflurane on Long-term Outcomes With Patients Undergoing Elective Excision of Primary Liver Tumors
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Tri-Service General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20220034
Record Dates: First submitted 2022-03-29; First posted 2022-04-18 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol Group (Experimental): The propofol group was maintained at an effect-site concentration (Ce) of 2.0-4.0 mcg/mL by a target-controlled infusion (TCI) system.
  Interventions: Drug: Propofol
- Sevoflurane group (Experimental): The sevoflurane group was maintained via sevoflurane vaporizer between 1% and 3% (target minimum alveolar concentration of 0.7-1.3 MAC).
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — total intravenous anesthesia with propofol for the partial hepatectomy of hepatocellular carcinoma.
  Other Names: total intravenous anesthesia
  Arms: Propofol Group
Drug: Sevoflurane — The sevoflurane group was maintained via sevoflurane vaporizer between 1% and 3% (target minimum alveolar concentration of 0.7-1.3 MAC).
  Arms: Sevoflurane group

SUMMARY:
This is a two-arm, parallel-group randomized clinical trial. Routine perioperative care would be performed in volunteers with primary Hepatocellular carcinoma. The study will enroll approximately 500 volunteers to compare the progression-free or overall survival in patients undergoing elective partial hepatectomy for primary liver tumors between propofol and sevoflurane for the maintenance of anesthesia.

DETAILED DESCRIPTION:
Before the scheduled procedure, the patients are randomly assigned into peopofol group or groups (1:1) according to the randomization generated by the computer. Both groups were induced with propofol 1~2.5 mg/kg propofol. The propofol group was maintained at an effect-site concentration of 2.0-4.0 mcg/mL by a target-controlled infusion system. The sevoflurane group was maintained via sevoflurane vaporizer between 1% and 3% (target minimum alveolar concentration of 0.7-1.3 MAC). During the operation, the dose of anesthetic drugs (propofol/fentanyl /remifentanil and sevoflurane/cisatracurium/rocuronium) are adjusted to maintain the mean arterial pressure and heartbeat fluctuations within 20% of the baseline value and Entropy (or BIS) value at 40-60in both groups. The following patient data were recorded, the type of anesthesia, sex, age at the time of surgery, preoperative Karnofsky performance status score and functional capacity, the postoperative complications within 30 days (according Clavien-Dindo classification), American Society of Anesthesiologists physical status scores, tumor size, intraoperative blood loss/transfusion, duration of surgery, duration of anesthesia, total opioid (remifentanil/fentanyl/ propofol) use, postoperative radiation therapy, postoperative chemotherapy, postoperative concurrent chemoradiotherapy, the presence of disease progression, and 6-month, 1-year, and 3-year overall survival and Karnofsky performance status score were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Twenty to eighty-year-old.
2. ASA class I-III.
3. Patients undergoing partial hepatectomy for hepatocellular carcinoma under general anesthesia.

Exclusion Criteria:

1. Severe mental disorder
2. Pregnant or lactating women
3. Morbidly obese
4. Allergy to any of the drugs used in this study
5. Recurrent tumor or repeat surgery
6. Biopsy cases
7. Incomplete data collection before the surgery
8. Palliative treatment after surgery
9. simultaneous treatment of other malignancies
10. Combined propofol and inhalation anesthesia or other anesthetics, such as ketamine or dexmedetomidine
11. Diagnosed as benign liver tumor
12. Emergency surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From the date of surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months"
  6-month overall survival, 1-year overall survival, and 3-year overall survival
The presence of disease progression | From the date of surgery until the date of first documented progression (recurrence or metastasis),assessed up to 36 months
  From the date of surgery until the date of first documented progression (recurrence or metastasis) or date of death from any cause, assessed up to 36 months"

SECONDARY OUTCOMES:
Postoperative complications | The period from the day of surgery to postoperative 30 days
  Clavien-Dindo classification, and other postoperative complications
Karnofsky performance status score | Karnofsky performance score(from 0 (dead) to 100(normal no complication)) before surgery (baseline data) , postoperation 7 days, postoperation 3 months, postoperation 6 months, postoperation 12 months
  to access patients' functional impairment
Length of hospital stays | from the day of surgery to dischage, assessed up to 30 days
  the length of stays in general ward and ICU

OTHER OUTCOMES:
time of operation and anesthesia | time of the total procedure
  record the time the operation and anesthesia
blood loss and blood transfusion | during the operation of partial hepatectomy
  record the blood loss (ml) and volume of blood transfusion (ml)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
depends the various challenges in this study.